CLINICAL TRIAL: NCT01612559
Title: A Registry Study on Safety Surveillance of Kudiezi (a Chinese Medicine Injection) Used in China
Brief Title: Safety Study of Kudiezi (a Chinese Medicine Injection) Used in Hospitals in China
Acronym: RSCMI-Ⅱ
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: China Academy of Chinese Medical Sciences (Other)
Collaborators: Dongfang Hospital Beijing University of Chinese Medicine (Other)
Responsible Party: Principal Investigator, Yanming Xie, Deputy Director, China Academy of Chinese Medical Sciences
Other Study IDs: RSCMI-Ⅱ; RSCMI-Ⅱ (Registry Identifier: Registry study on Chinese Medicine Injection)
Record Dates: First submitted 2012-06-03; First posted 2012-06-06 (Estimated); Last update posted 2012-06-06 (Estimated); Status verified 2012-06

CONDITIONS: Coronary Heart Disease; Angina Pectoris
MeSH Terms: conditions — Coronary Disease; Angina Pectoris

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
This study was advocated by Institute of Basic Research in Clinical Medicine, China Academy of Chinese Medical Sciences in October 2011.

It was funded by China major scientific and technological specialized project for 'significant new formulation of new drugs'.

Kudiezi is kind of Chinese Medicine injection used for treating coronary heart disease and angina pectoris in many Chinese hospitals.

The purpose of this study is to determine adverse drug events or adverse drug reaction in large sample size 30,000 patients.

DETAILED DESCRIPTION:
It is very common that Chinese Medicine Injection used in hospitals in mainland China. However safety problems rose in recent years. There could be many uncertain factors influence Chinese Medicine Injection in clinical practice.

Safety surveillance on Chinese Medicine injection is an important problem that needs to be sorted out through large sample observational study.

A registry study for Kudiezi injection safety surveillance with 30000 patients will be conducted from Jan.2012 to Dec.2015.

Eligibility criteria Patients who will use Kudiezi injection in selected hospitals

Data will be collected in four aspects by four different forms as following:

Form A (blue): demographic information Form B (yellow): adverse drug events/reaction Form C (white): extracted information from hospital information system and laboratory information system Form D (red): personalized information

ELIGIBILITY:
Inclusion Criteria:

* Patients using Kudiezi injection from 2012 to 2014

Exclusion Criteria:

* none

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: An anticipated sample size was caculated in this study, about 30000. Patients using Kudiezi injection from 2012 to 2014 in more than 20 hospitals.
Sampling Method: Non-Probability Sample
Enrollment: 30000 (Estimated)
Dates: Start 2012-01; Primary Completion 2014-12 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Number of participants with adverse events; incidence of Kudiezi'ADRs and identify factors that contributed to the occurrence of the adverse reaction | to assess Kudiezi's 'adverse event' and 'drug adverse reaction' during patients' hospital stay, administration information of Kudiezi will be registered every day. The registry procedure will last 3 years only for patients using Kudiezi.
  All patients will be measured and assessed at the time Kudiezi is administered to them until they discharge. Patients using Kudiezi will be registered on a registration form including disease background, Kudiezi's administration, and extraction information from hospital information system. An adverse event or drug adverse reaction form also will be used to describe any doubted symptoms or signs from patients. A judgment will be made by doctors directly and a further analysis will be conducted by researchers to decide those potential side effects of Kudiezi.

CONTACTS AND LOCATIONS:
Overall Officials: Yan M Xie, BA, Principal Investigator — Institute of Basic Research in Clinical Medicine, China Academy of Chinese Medical Sciences